CLINICAL TRIAL: NCT06296472
Title: De Quervain's Disease in the Acute Phase: Randomized Interventional Study Aimed at Evaluating the Effectiveness of Standard Physiotherapy Treatment (HANDGUIDE), Compared to Experimental Treatment After Performing Ultrasound-guided Infiltrative Therapy.
Brief Title: De Quervain's Disease in the Acute Phase:a Study Aimed at Evaluating the Effectiveness of Standard Physiotherapy Treatment (HANDGUIDE), Compared to Experimental Treatment After Performing Ultrasound-guided Infiltrative Therapy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDQ23
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: De Quervain Disease; Hand Tenosynovitis
Keywords: Hand rehabilitation
MeSH Terms: conditions — De Quervain Disease | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator)
  Interventions: Other: Standard
- Experimental (Experimental)
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — -the experimental group will carry out a program of eccentric exercises following the infiltration and will also wear the wrist brace for 4 weeks.
  Arms: Experimental
Other: Standard — -the standard group will carry out a program of generic exercises following the infiltration and will also wear the wrist brace for 4 weeks.
  Arms: Standard

SUMMARY:
The objective of the study is to compare pain reduction and disability reduction in two groups of patients diagnosed with de Quervain syndrome who will undergo ultrasound-guided infiltrative treatment with corticosteroid as per normal clinical practice:

* the control group will subsequently be subjected to a standard treatment based on the European guidelines of the HANDGUIDE group,
* the experimental group will subsequently carry out a program of eccentric exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with a minimum age of 18 years;
* Medical diagnosis of de Quervain syndrome assessed through orthopedic clinical examination e confirmation by ultrasound;
* Signing of the informed consent and participation in the study.

Exclusion Criteria:

* Patients who are not self-sufficient or not able to understand and want;
* Presence of other pathologies in the hand affected by de Quervain pathology, such as intersection syndrome, neuropathies, fractures, rhizoarthrosis, arthrosis of the radio-carpal or intercarpal joint, intercarpal instability, cervical radiculopathy, rheumatic or metabolic pathologies;
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | At baseline (day 0)
  An 11-point Numeric Pain Rating Scale (NPRS) ranging from 0 to 10 was anchored on the left with the phrase "No Pain" and on the right with the phrase "Worst Imaginable Pain." Patients rated their current, best, and worst level of pain during the last 24 hours.
Numeric Pain Rating Scale | After 1 month
  An 11-point Numeric Pain Rating Scale (NPRS) ranging from 0 to 10 was anchored on the left with the phrase "No Pain" and on the right with the phrase "Worst Imaginable Pain." Patients rated their current, best, and worst level of pain during the last 24 hours.
Numeric Pain Rating Scale | After 3 months
  An 11-point Numeric Pain Rating Scale (NPRS) ranging from 0 to 10 was anchored on the left with the phrase "No Pain" and on the right with the phrase "Worst Imaginable Pain." Patients rated their current, best, and worst level of pain during the last 24 hours.
Numeric Pain Rating Scale | After 6 months
  An 11-point Numeric Pain Rating Scale (NPRS) ranging from 0 to 10 was anchored on the left with the phrase "No Pain" and on the right with the phrase "Worst Imaginable Pain." Patients rated their current, best, and worst level of pain during the last 24 hours.

SECONDARY OUTCOMES:
Disabilities of Arm, Shoulder and Hand | At baseline (day 0)
  The Disabilities of Arm, Shoulder and Hand (DASH) score consists of 30 questions and is used to assess functional disorders of the upper extremity. The possible score ranges from 0 to 100 points. 0 points represent a complete, unrestricted function of the upper extremities, while 100 points represent the greatest possible functional impairment.
Disabilities of Arm, Shoulder and Hand | After 1 month
  The Disabilities of Arm, Shoulder and Hand (DASH) score consists of 30 questions and is used to assess functional disorders of the upper extremity. The possible score ranges from 0 to 100 points. 0 points represent a complete, unrestricted function of the upper extremities, while 100 points represent the greatest possible functional impairment.
Disabilities of Arm, Shoulder and Hand | After 3 months
  The Disabilities of Arm, Shoulder and Hand (DASH) score consists of 30 questions and is used to assess functional disorders of the upper extremity. The possible score ranges from 0 to 100 points. 0 points represent a complete, unrestricted function of the upper extremities, while 100 points represent the greatest possible functional impairment.
Disabilities of Arm, Shoulder and Hand | After 6 months
  The Disabilities of Arm, Shoulder and Hand (DASH) score consists of 30 questions and is used to assess functional disorders of the upper extremity. The possible score ranges from 0 to 100 points. 0 points represent a complete, unrestricted function of the upper extremities, while 100 points represent the greatest possible functional impairment.
Patient-Rated Wrist Evaluation | At baseline (day 0)
  The Patient-Rated Wrist Evaluation (PRWE) is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living.
Patient-Rated Wrist Evaluation | After 1 month
  The Patient-Rated Wrist Evaluation (PRWE) is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living.
Patient-Rated Wrist Evaluation | After 3 months
  The Patient-Rated Wrist Evaluation (PRWE) is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living.
Patient-Rated Wrist Evaluation | After 6 months
  The Patient-Rated Wrist Evaluation (PRWE) is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Wolf JM, Sturdivant RX, Owens BD. Incidence of de Quervain's tenosynovitis in a young, active population. J Hand Surg Am. 2009 Jan;34(1):112-5. doi: 10.1016/j.jhsa.2008.08.020. Epub 2008 Dec 10. PMID 19081683
- [Result] Walker-Bone K, Palmer KT, Reading I, Coggon D, Cooper C. Prevalence and impact of musculoskeletal disorders of the upper limb in the general population. Arthritis Rheum. 2004 Aug 15;51(4):642-51. doi: 10.1002/art.20535. PMID 15334439
- [Result] Ferrara PE, Codazza S, Cerulli S, Maccauro G, Ferriero G, Ronconi G. Physical modalities for the conservative treatment of wrist and hand's tenosynovitis: A systematic review. Semin Arthritis Rheum. 2020 Dec;50(6):1280-1290. doi: 10.1016/j.semarthrit.2020.08.006. Epub 2020 Aug 29. PMID 33065423